CLINICAL TRIAL: NCT00673491
Title: Diffusion of Clinical Pathways for the Implementation of Effective and Appropriate Care
Brief Title: Clinical Pathways for Effective and Appropriate Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agenzia Regionale Sanitaria delle Marche (Other Government)
Collaborators: Agenzia Nazionale per i Servizi Sanitari Regionali (Other); Regione Friuli Venezia Giulia (Unknown); Reggio Calabria (Other); Forum della Solidarieta (Unknown); IRCCS Besta (Unknown); Regione Molise (Unknown); Regione Puglia (Unknown); Regione Siciliana (Unknown); Regione Umbria (Unknown); University of Eastern Piedmont (Other)
Responsible Party: Andrea Gardini, Agenzia Regionale Sanitaria delle Marche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DCPIEAC-EXART12MARCHE
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-05

CONDITIONS: Stroke
Keywords: Critical Pathways; Stroke; Randomized Controlled Trial; Effectiveness
MeSH Terms: conditions — Stroke | interventions — Critical Pathways

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients treated according to clinical pathways
  Interventions: Other: Clinical Pathways
- 2 (No Intervention): Patients treated according to usual care

INTERVENTIONS:
Other: Clinical Pathways — Clinical pathways are a methodology for the mutual decision making and organization of care for a well-defined group of patients during a well-defined period. Defining characteristics of clinical pathways includes: an explicit statement of the goals and key elements of care based on evidence, best practice, and patient expectations; the facilitation of the communication, coordination of roles, and sequencing the activities of the multidisciplinary care team, patients and their relatives; the documentation, monitoring, and evaluation of variances and outcomes; and the identification of the appropriate resources.
  Arms: 1

SUMMARY:
The purposes of this study are to determine whether clinical pathways: 1)improve the quality of the care provided to patients affected by stroke in terms of clinical outcomes, efficiency continuity of care and patients' satisfaction; 2) facilitate the use of evidence based medicine in clinical practice.

DETAILED DESCRIPTION:
The coordination of care has been proved to be able to improve prognosis in acute stroke patients. Prompt identification of symptoms, organised timely and efficient transportation towards appropriate facilities, has become essential part of effective treatment, as well as organized rehabilitation. The importance of organized stroke care in facilitating recovery has been recognized for the last 10 years, but it is still unclear how organized care contributes to improved outcomes. Since clinical pathways aim to promote evidence- and guideline-based care, improve the organisation and efficiency of care, and reduce cost, their implementation may be a method for achieving the organizational standards required to grant appropriate care in stroke. Even though in the past decade, care pathways have been increasingly implemented as a tool in acute stroke care and stroke rehabilitation the evidence supports partially the use of clinical pathways in stroke because very little prospective controlled data demonstrated their effectiveness through the continuum of the care. Our study was designed in order to conduct a rigorous evaluation of clinical pathways for treatment of acute stroke patients in different types of organized stroke care.

ELIGIBILITY:
Inclusion Criteria:

* Principal diagnosis of Ischemic Stroke (ICD9CM code 434.91)

Exclusion Criteria:

* Transient cerebral ischemia (ICD9CM code 435.9)
* Intracerebral hemorrhage (ICD9CM codes 431.xx)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2005-07; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days after hospital admission

SECONDARY OUTCOMES:
Disability | At hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Di Stanislao, MD, Study Chair — Agenzia Regionale Sanitaria delle Marche

REFERENCES:
- [Derived] Panella M, Marchisio S, Brambilla R, Vanhaecht K, Di Stanislao F. A cluster randomized trial to assess the effect of clinical pathways for patients with stroke: results of the clinical pathways for effective and appropriate care study. BMC Med. 2012 Jul 10;10:71. doi: 10.1186/1741-7015-10-71. PMID 22781160
- [Derived] Panella M, Marchisio S, Barbieri A, Di Stanislao F. A cluster randomized trial to assess the impact of clinical pathways for patients with stroke: rationale and design of the Clinical Pathways for Effective and Appropriate Care Study [NCT00673491]. BMC Health Serv Res. 2008 Nov 3;8:223. doi: 10.1186/1472-6963-8-223. PMID 18980664